CLINICAL TRIAL: NCT06141824
Title: Performance Evaluation of the Lucira COVID-19 & Flu Test Versus FDA Authorized SARS-CoV-2 and Influenza A&B Assays
Brief Title: Performance Evaluation of the Lucira COVID-19 & Flu Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucira Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09A-CLI-001
Record Dates: First submitted 2023-08-03; First posted 2023-11-21 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Influenza
Keywords: COVID-19; Influenza; COVID-19 test; Multiplex test; RT-LAMP; Molecular test; Single-use test
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Subject Self-Collection and Specimen Testing (Experimental): A subject's participation in this study will consist of one study visit. The subject self-collects a nasal swab sample according to Lucira COVID- 19 & Flu Test instructions and runs test according to QRI.
  Following the Lucira COVID-19 & Flu Test self-collection will be an additional swab collection for reference method testing. One (1) additional NS specimen will be collected by the healthcare professional, prepared in Transport Medium, and sent to the reference laboratory.
  Interventions: Device: Lucira COVID-19 & Flu Test

INTERVENTIONS:
Device: Lucira COVID-19 & Flu Test — The Lucira COVID-19 & Flu Test is a rapid, single-use, molecular test for the qualitative detection and discrimination of SARS-CoV-2, Influenza A, and Influenza B viral RNA in nasal swab samples.

SUMMARY:
The Lucira COVID-19& Flu Test is a single use (disposable) RT-LAMP test kit intended for the simultaneous rapid in vitro qualitative detection and differentiation of SARS-CoV-2, Influenza A, and Influenza B viral RNA in anterior nasal swab specimens.

The test consists of a nasal swab, a sample vial the nasal swab sample is placed in the sample vial, containing the sample buffer, and the test unit, which detects whether SARS-CoV-2, Influenza A, and Influenza B virus is present within the specimen during an acute infection. The Lucira test uses a proprietary, molecular based process to detect the presence of SARS-CoV-2, Influenza A, or Influenza B virus. The purpose of this study is to investigate the Lucira COVID-19 & Flu Test for the in vitro qualitative detection and differentiation of RNA from SARS-CoV-2, Influenza A, and Influenza B in nasal swab specimens from patients suspected of COVID-19 or Influenza A or Influenza B. The primary objective is to test at least 1000 self-collected nasal swab samples and to confirm the Lucira COVID-19 & Flu Test provides similar accuracy to a high complexity lab molecular diagnostic RT-PCR assay(s) with known high sensitivity for detecting SARS-CoV-2, Influenza A, and Influenza B virus.

DETAILED DESCRIPTION:
The study is a prospective study with seven (7) sites in the U.S. participating in the study. The Investigational device was tested on-site, and the comparator samples were sent to reference laboratories in the U.S. Reference testing was performed by trained laboratory personnel. This investigational device testing was performed in a simulated-home environment with medical staff on site and included nasal swabs self-collected by study subjects per the quick reference instructions (QRI).

A qualified research person was designated as the Investigator at each site with the responsibility for oversight of the study in accordance with Good Clinical Practice (GCP) and regulatory requirements.

The protocol and subject informed consent were reviewed by an Institutional Review Board (IRB) and written IRB approval was issued prior to enrollment of subjects into the study at that site.

A subject's participation in this study consisted of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject then received a unique study identification number. Subject demographics including age, sex, race, ethnicity, education level, employment status, and income was also collected at that time.

Two (2) swabs were collected for this study: One (1) nasal swab for the Lucira COVID-19 & Flu Test and one (1) nasal swab for reference testing. These two study swabs were both collected similarly as directed in the Lucira COVID-19 & Flu Test QRI. Any swab specimens required for routine standard of care testing were collected prior to the specimens collected for this investigation.

Subjects aged 14 years or older self-collected a nasal swab sample and ran the Lucira COVID-19 Test according to QRI in the test kit. Nasal swab sample collection and testing for Subjects ≥ 2 years but <14 years of age was assisted by a subject meeting the requirement for self-collection. The subject was observed during the swabbing collection by the HCP and HCP documented collection details and any collection issues. Nasal swabs obtained from self-collection were discarded after having been used for testing per QRI. HCP interpreted and documented results.

Following the Lucira COVID-19 Test self-collection an additional swab was collected for reference method testing. One (1) additional NS specimen was collected by the health care professional, prepared in Transport Medium, and sent for reference laboratory testing. Each collection, the Lucira swab and reference swab, had a potential maximum of two swabs, including retests, for a maximum of four swabs per visit.

Reference labs received study sample aliquots and tested samples against FDA emergency use authorized SARS-CoV-2 and FDA cleared Influenza A&B Assays. Reference testing characterized specimens as negative or positive for SARS-CoV-2 and Influenza A&B. Therefore, positive percent agreement (PPA) and negative percent agreement (NPA) of the Lucira COVID-19 & Flu Test was calculated by comparison with the respective reference methods.

Additional testing on remaining remnant aliquots may be performed to investigate any discrepant and discordant results as needed by other FDA cleared/authorized molecular methods.

At the end of the study, and at the Sponsor's discretion, residual remnant aliquots shall remain at the reference laboratory, be destroyed/discarded, or returned to the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 14 years and older (self-collected) or individuals less than 14 years old but ≥ 2 years old (collected by an adult)
* Human subjects suspected of respiratory viral infection consistent with COVID-19 or Influenza by their healthcare provider within 4 days of symptom onset
* Must be willing to try Lucira COVID-19 & Flu test with an anterior nasal (nasal) swab specimen collected from both nostrils
* Subject information shall include: gender, age, collection date, collection time, race, ethnicity, temperature, signs/symptoms, date of symptom onset, symptom severity, vaccination status, household income, education status, employment status, routine test data (results, methodology, date of collection, if available)

Exclusion Criteria:

* Currently suffering from nasal trauma such as a nosebleed
* Received a nasal rinse/wash/aspirates for standard of care testing
* The subject is undergoing treatment for COVID-19 or Flu currently and/or within the past 14 days of the study visit, including but not limited to: inhaled influenza vaccine (FluMist®) or flu antiviral medication, which may include but is not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), or Baloxavir marboxil (Xofluza®).
* The subject is currently receiving or has received within the past 30 days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
* The subject has previously participated in this research study
* Incorrect comparator swab type or transport media
* Incorrect specimen handling
* Subjects not consented

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1361 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cullman Clinical Trials, Cullman, Alabama
  - Benchmark Research, Colton, California
  - Carbon Health, Oakland, California
  - Koch Family Medicine, Morton, Illinois
  - Lakeside Life Science, Plymouth, New Hampshire
  - Carbon Health, Eatontown, New Jersey
  - Benchmark Research, San Angelo, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1366 research participants were consented to participate in the study, 5 participants were withdrawn from the study. 1361 participants were enrolled and participated in the study.
Groups:
- Lucira COVID-19 & Flu Test: The Lucira COVID-19 (Coronavirus 2019) and Flu Test is a rapid, single-use, molecular test for the qualitative detection and discrimination of SARS-CoV-2, Influenza A, and Influenza B viral RNA in nasal swab samples. Participants self-collected an anterior nasal swab sample.
Period: Overall Study
Arm/Group | Lucira COVID-19 & Flu Test
Started | 1361
Evaluable COVID-19 Results | 1229
Evaluable Flu A Results | 1333
Evaluable Flu B Results | 1332
Completed | 1361
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 1361 subjects enrolled, 1229 had evaluable COVID-19 results, 1333 had evaluable Flu A results and 1332 had evaluable Flu B results. The population used for analysis is enrolled participants. Data is presented for participants who took test for COVID-19, Flu A and Flu B.
Arm/Group | Lucira COVID-19 & Flu Test
Number analyzed (Participants) | 1361
Age, Customized [Count of Participants; unit: Participants] — Population: "Overall Number of Participants" signifies participants evaluable for COVID-19, Flu A and Flu B results respectively. "Number Analyzed" signifies number of participants evaluable for specified rows.
  Participants
    COVID-19: number analyzed (Participants) | 1229
    COVID-19: 2-5 years | 48
    COVID-19: 6-21 years | 342
    COVID-19: 22-59 years | 708
    COVID-19: >=60 years | 131
    Flu A: number analyzed (Participants) | 1333
    Flu A: 2-5 years | 52
    Flu A: 6-21 years | 377
    Flu A: 22-59 years | 763
    Flu A: >=60 years | 141
    Flu B: number analyzed (Participants) | 1332
    Flu B: 2-5 years | 52
    Flu B: 6-21 years | 376
    Flu B: 22-59 years | 763
    Flu B: >=60 years | 141
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: "Overall Number of Participants" signifies participants evaluable for COVID-19, Flu A and Flu B results respectively. "Number Analyzed" signifies number of participants evaluable for specified rows.
  Participants
    COVID-19: number analyzed (Participants) | 1229
    COVID-19: Female | 763
    COVID-19: Male | 465
    COVID-19: Other | 1
    Flu A: number analyzed (Participants) | 1333
    Flu A: Female | 834
    Flu A: Male | 498
    Flu A: Other | 1
    Flu B: number analyzed (Participants) | 1332
    Flu B: Female | 834
    Flu B: Male | 497
    Flu B: Other | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: "Overall Number of Participants" signifies participants evaluable for COVID-19, Flu A and Flu B results respectively. "Number Analyzed" signifies number of participants evaluable for specified rows.
  Participants
    COVID-19: number analyzed (Participants) | 1229
    COVID-19: Hispanic or Latino | 262
    COVID-19: Not Hispanic or Latino | 955
    COVID-19: Unknown or Not Reported | 12
    Flu A: number analyzed (Participants) | 1333
    Flu A: Hispanic or Latino | 271
    Flu A: Not Hispanic or Latino | 1044
    Flu A: Unknown or Not Reported | 18
    Flu B: number analyzed (Participants) | 1332
    Flu B: Hispanic or Latino | 271
    Flu B: Not Hispanic or Latino | 1043
    Flu B: Unknown or Not Reported | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Overall Number of Participants" signifies participants evaluable for COVID-19, Flu A and Flu B results respectively. "Number Analyzed" signifies number of participants evaluable for specified rows.
  Participants
    COVID-19: number analyzed (Participants) | 1229
    COVID-19: American Indian or Alaska Native | 2
    COVID-19: Asian | 16
    COVID-19: Native Hawaiian or Other Pacific Islander | 2
    COVID-19: Black or African American | 57
    COVID-19: White | 1112
    COVID-19: Other | 25
    COVID-19: Unknown or Not Reported | 15
    Flu A: number analyzed (Participants) | 1333
    Flu A: American Indian or Alaska Native | 2
    Flu A: Asian | 18
    Flu A: Native Hawaiian or Other Pacific Islander | 2
    Flu A: Black or African American | 62
    Flu A: White | 1206
    Flu A: Other | 28
    Flu A: Unknown or Not Reported | 15
    Flu B: number analyzed (Participants) | 1332
    Flu B: American Indian or Alaska Native | 2
    Flu B: Asian | 18
    Flu B: Native Hawaiian or Other Pacific Islander | 2
    Flu B: Black or African American | 62
    Flu B: White | 1205
    Flu B: Other | 28
    Flu B: Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Confirmation That the Lucira COVID-19 & Flu Test Provides Similar Performance to a High Complexity Lab Molecular Diagnostic RT-PCR Assay(s) With Known High Sensitivity
Description: The sensitivity and specificity endpoint are Percent Positive Agreement (PPA) ≥80%/Negative Positive Assessment (NPA) ≥98% for COVID-19 and PPA ≥90%/NPA ≥95% for Flu A&B as compared to FDA emergency use authorized SARS-CoV-2 and FDA cleared Influenza A+B Assays. Two (2) swabs were collected for this study: One (1) anterior nasal swab (NS) for the Lucira COVID-19 and Flu Test and one (1) NS for reference testing. Reference testing characterized specimens as negative or positive for SARS-CoV-2 and Influenza A and B. Therefore, PPA and NPA of the Lucira COVID-19 and Flu Test were calculated by comparison with the respective reference methods. The data were analyzed via comparison to the comparator method in this protocol in a standard 2x2 table, with PPA and NPA calculated against the comparator. The percentage of the expected result was computed individually along with the associated 95% Wilson Score Confidence Interval [1] for each panel.
Time Frame: Day 1
Population: "Overall Number of Participants" signifies participants evaluable for COVID-19, Flu A and Flu B results respectively. "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of results matching PCR
Groups:
- COVID-19: Participants who were evaluable for COVID-19 results.
- Flu A: Participants who were evaluable for Flu A results.
- Flu B: Participants who were evaluable for Flu B results.
Arm/Group | COVID-19 | Flu A | Flu B
Number analyzed (Participants) | 1229 | 1333 | 1332
percentage of results matching PCR
  Percent Positive Agreement (PPA): number analyzed (Participants) | 141 | 123 | 0
  Percent Positive Agreement (PPA) | 88.7 [82.4 to 92.9] | 90.2 [83.7 to 94.3] |
  Negative Positive Agreement (PPA): number analyzed (Participants) | 1088 | 1210 | 1332
  Negative Positive Agreement (PPA) | 99.7 [99.2 to 99.9] | 99.4 [98.8 to 99.7] | 99.9 [99.6 to 100.0]

ADVERSE EVENTS:
Time Frame: From the time of the beginning of enrollment to study completion, which was approximately 16 weeks.
Groups:
- Lucira COVID-19 & Flu Test: The Lucira COVID-19 & Flu Test is a rapid, single-use, molecular test for the qualitative detection and discrimination of SARS-CoV-2, Influenza A and Influenza B viral RNA in nasal swab samples.
Arm/Group | Lucira COVID-19 & Flu Test
All-Cause Mortality (participants affected / at risk) | 0/1361
Serious Adverse Events (participants affected / at risk) | 0/1361
Other Adverse Events (participants affected / at risk) | 0/1361

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT06141824/Prot_SAP_000.pdf